CLINICAL TRIAL: NCT02863406
Title: MINASARC01: Comparison of Characteristics of Bronchoalveolar Lavage Dusting and of Specific Questionnary Data in Healthy Volunteers and Patients Suffering From Sarcoidosis: Pilot Study, Prospective, Multicenter, Multidisciplinary With Blind Analysis
Brief Title: Comparison of Characteristics of Bronchoalveolar Lavage Dusting and of Specific Questionnary Data in Healthy Volunteers and Patients Suffering From Sarcoidosis
Acronym: MINASARC01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Collaborators: Sciences Po Paris (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MINASARC01
Record Dates: First submitted 2016-07-05; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Sarcoidosis
Keywords: Dust rate; Microscopic analysis
MeSH Terms: conditions — Sarcoidosis | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Experimental): Bronchoalveolar lavage in healthy volunteers
  Interventions: Other: Bronchoalveolar lavage
- Patients suffering from sarcoidosis (Experimental): Bronchoalveolar lavage in patients suffering from sarcoidosis
  Interventions: Other: Bronchoalveolar lavage

INTERVENTIONS:
Other: Bronchoalveolar lavage — Bronchoalveolar lavage in order to determine rate of dust

SUMMARY:
Comparison of dusting rate of bronchoalveolar lavage in healthy volunteers and patients suffering from sarcoidosis.

Blind analysis of bronchoalveolar lavage with Optical Microscopy, Transmission Electron Microscopy and MicroAnalysis.

For patients, comparison of bronchoalveolar lavage, pathological examination of biopsies (Optical Microscopy, Transmission Electron Microscopy and MicroAnalysis) and specific Professional and environmental questionnary.

Healthy volunteers matched with patients regarding to age (every 10 years), sex and tobacco consumption (non-smoking, smoking less than 5 pack-year, smoking between 5 and 10 pack-year, smoking more than 10 pack-year)

ELIGIBILITY:
Inclusion Criteria:

* Absence of respiratory and cardiac illness (healthy volunteers)
* Normal spirometry and chest x-ray (healthy volunteers)
* Absence of viral infection (B and C hepatitis, HIV) (healthy volunteers)
* Confirmation of sarcoidosis (endoscopic exam with bronchoalveolar lavage) (patients suffering from sarcoidosis)

Exclusion Criteria:

* Pregnant women
* Lack of bronchoalveolar lavage (volume less than 20 ml)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Significant difference between dusting rate of bronchoalveolar lavage in healthy volunteers and patients suffering from sarcoidosis (analysis by Optical Microscopy, Transmission Electron Microscopy and MicroAnalysis). | Procedure of bronchoalveolar lavage

SECONDARY OUTCOMES:
Correlation between mineral overload of bronchoalveolar lavage for patient suffering from sarcoidosis and data extracted from specific Professional and environmental questionnary | Through study completion, an average of 1 year
Correlation between mineral overload of bronchoalveolar lavage for patient suffering from sarcoidosis and pathological examination of biopsies (analysis by Optical Microscopy, Transmission Electron Microscopy and MicroAnalysis). | Through study completion, an average of 1 year
Interest of macrophagic dusting index | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michel Vincent, MD, Principal Investigator — Centre Hospitalier Saint Joseph Saint Luc

IPD SHARING:
Plan to Share IPD: No